CLINICAL TRIAL: NCT05905614
Title: An Open-label, Dose-escalation, Phase I Clinical Trial to Explore the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SPH4336 Tablets in the Treatment of Advanced Solid Tumors
Brief Title: Phase I Clinical Study of SPH4336 Tablets in the Treatment of Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH4336-101
Record Dates: First submitted 2023-05-29; First posted 2023-06-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH4336 Tablets (Experimental): SPH4336 Tablets
  Interventions: Drug: SPH4336 Tablets

INTERVENTIONS:
Drug: SPH4336 Tablets — Open-label SPH4336 Tablets ：Administered by oral

SUMMARY:
This clinical study evaluated the safety and efficacy of SPH4336 in the treatment of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced solid tumors；
2. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1；
3. Life expectancy ≥ 3 months；
4. Good organ function；
5. According to the investigator's judgment, the patient could comply with the trial protocol;
6. Patients who voluntarily participate in this study, completely understand this study, and voluntarily sign the informed consent form (ICF).

Exclusion Criteria:

1. Received other antineoplastic therapy before the first dose；
2. Had a major surgery before the first dose of study medication or was planned to have a major surgery after starting the study medication;
3. Enroll in other clinical trials and receive treatment as a subject before initial medication;
4. Patients with allergic constitution or history of severe allergy;
5. Hepatitis B surface antigen [HBsAg] positive and HBV-DNA copy number ≥500 copies /ml or 100 IU/ml, HCV-Ab positive and HCV-RNA higher than the detection limit of the research center; A history of immunodeficiency;
6. Cardiac criteria: presence of factors that may cause QTc prolongation or arrhythmia such as congestive heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, and other concomitant medications known to prolong the QT interval. The presence of any unstable cardiovascular disease;
7. Hypertension that cannot be effectively controlled after treatment;
8. Have severe lung disease;
9. Pregnant and lactating women;
10. Female patients of reproductive age and male patients with a partner of reproductive age who were unwilling to use effective contraception throughout the trial;
11. Concomitant diseases that seriously endanger patient safety or affect the completion of the study according to the investigator's judgment;
12. Had a definite history of neurological or mental disorders;
13. Other circumstances considered by the investigator to be inappropriate for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose（MTD） | Up to 28 days
  Measurement of MTD of SPH4336 in all subjects
Dose-limiting toxicity (DLT) | Up to 28 days
  Measurement of DLT of SPH4336 in all subjects

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
Progression-free survival (PFS) | Up to 1 year
  From the start date of study treatment to the date of progression disease or death , whichever occurred first.
Cmax | predose,1,2,4,5,6,8,10,12,24 hours post-dose
  PK (Pharmacokinetics) parameters
Tmax | predose,1,2,4,5,6,8,10,12,24 hours post-dose
  PK (Pharmacokinetics) parameters
Disease control rate (DCR) | Up to 1 year
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease.
Duration of remission (DOR) | Up to 1 year
  DOR was defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response to the date of disease progression per RECIST v1.1 or death from any cause.
Safety and tolerability | Up to 1 year
  Adverse event type, incidence, duration, correlation with study drug.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Jinan Central Hospital, Jinan, Shandong
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Peking University Cancer Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing

REFERENCES:
- [Derived] Jiang Y, Liang X, Sun ML, Gao G, Gong Y, Li HP, Liu J, Wang YS. Phase I trial of SPH4336, a novel cyclin-dependent kinase 4/6 inhibitor, in patients with advanced solid tumors. Oncologist. 2025 Jun 4;30(6):oyaf077. doi: 10.1093/oncolo/oyaf077. PMID 40586764